CLINICAL TRIAL: NCT04935970
Title: Metabolic Disorders and Their Correction in Vertigo and Unsteadiness
Brief Title: Metabolic Disorders and Vertigo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 16-19
Record Dates: First submitted 2021-04-11; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-03

CONDITIONS: Benign Paroxysmal Positional Vertigo (BPPV); Vestibular Migraine; Central Positional Vertigo; Vestibular Neuritis; Meniere Disease
Keywords: Benign paroxysmal positional vertigo (BPPV); vestibular neuritis; vestibular migraine; central positional vertigo; Meniere disease; persistent postural-perceptual dizziness (PPPD); vitamin D deficiency; hyperhomocysteinaemia
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vestibular Neuronitis; Meniere Disease; Vitamin D Deficiency; Hyperhomocysteinemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with peripherial vestibular disorder: Forty patients with BPPV, vestibular neuritis or another peripherial vestibular disorder
  Interventions: Diagnostic Test: diagnostic blood test; Diagnostic Test: neuropsychological test
- patients with central vestibular disorder: Forty patients vestibular disorder of central origin
  Interventions: Diagnostic Test: diagnostic blood test; Diagnostic Test: neuropsychological test
- healthy controls: twenty healthy control without balance problems
  Interventions: Diagnostic Test: diagnostic blood test

INTERVENTIONS:
Diagnostic Test: diagnostic blood test — vitamin D deficiency/insufficiency reveal, hyperhomocysteinaemia reveal
Diagnostic Test: neuropsychological test — neuropsychological test, including tas-26 scale, Beck's Depression Inventory, Spielberg-Hanin'scale.
  Groups: patients with central vestibular disorder; patients with peripherial vestibular disorder

SUMMARY:
The purpose of investigation is to assess the levels of metabolic factors (hydroxyvitamin D, homocysteine) between patients with vestibular dysfunction of peripheral origin (BPPV) and central origin (vestibular migraine). Also we will analyse another factors (such as anxiety and depression) and optimize therapeuthical approach accordingly with the data.

DETAILED DESCRIPTION:
Dizziness causes up to 2 to 15% of primary neurological complaints. In some patients who have undergone acute vertigo, postural instability, persistent postural perceptual vertigo (PPPV) develops, while in other similar cases occurs full recovery. So, it is necessary to search for neurophysiological, metabolic and psychophysiological factors and associated premorbid conditions that affect the outcome of neurovestibular compensation.

The case-control study will include 2 groups of patients suffering from vertigo of central and peripherial etiology. First group is recruited with patients were diagnosed with peripherial vestibular disorders, such as benign paroxysmal positional vertigo (BPPV), Meniere disease, vestibular neuritis. The proposal number of subjects in the first group is about forty. The second group will consist of forty patients with central vestibular disfunction: vestibular migraine, central positional vertigo etc. The inclusion of patient with persistent postural perceptual dizziness is discussed. Patients will be tested for hydroxyvitamin D and homocysteine in serum using an enzyme-linked immunosorbent assay (ELISA). The perception of the severity of disability was assessed using the Dizziness scale Handicap Inventory (DHI). All patients will undergo psychological test, including tas-26 scale, Beck's Depression Inventory, Spielberg-Hanin'sscale. Statistical analysis was carried out with the Statistical Analysis System (SAS) package. The relationships will be assessed using the chi squared test and logistic regression. The level of significance is set at p < 0.05. The methods for small samples (Mann-Whitney U ) will be used. It is presumed that differences in vitamin D levels beetween two groups will be considerable.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of participation in the study;
* Age:over 18 years old
* complaints of dizziness and insteadiness

Exclusion Criteria:

* Severe cognitive impairment (dementia)
* Severe depression
* Syncopal paroxysms
* Epileptic seizures
* Orthostatic hypotension
* Severe arrhythmia, unstable angina pectoris, acute myocardial infarction
* Pregnancy 8. Alcoholism, substance abuse and drug addiction
* Organic liver and kidney diseases with the development of functional disorders.
* Anemia (hemoglobin <10.5 g / dl for women and <11.5 g / dl for men)
* Active oncological process
* Demyelinating and neurodegenerative diseases.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients from clinic with damage of peripheral and central origin
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
vitamin D deficiency/insufficiency reveal | Through 1-6 months of diagnosis established.
  enzyme-linked immunosorbent assay (ELISA).
hyperhomocysteinaemia reveal | Through 1-6 months of diagnosis established.
  enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
correlation between metabolic and neuropsychological disorders | through study completion, an average of 1 year
  neuropsychological test, including tas-26 scale, Beck's Depression Inventory, Spielberg-Hanin'scale.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Bedenko, PhD student, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- Clinic of Neurology and Neurosurgery of I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
I give my consent to provide actual study protocol. However, It is impossible to provide stastistical documents and primary patient's documentation (It is forbidden by Local Ethic Committee of Sechenov University)

REFERENCES:
- [Background] Bedenko A.S., Antonenko L.М., Barinov A.N. Metabolic disorders in the pathogenesis of various causes of dizziness and instability // Annals of the Russian academy of medical sciences. - 2020. - Vol. 75. - N. 6. - P. 605-608. doi: 10.15690/vramn1244
- [Background] Bedenko A.S. Vertigo in neurological practice: rare causes and difficult decisions. Medical alphabet. 2019;2(19):34-36. (In Russ.) https://doi.org/10.33667/2078-5631-2019-2-19(394)-34-36
- [Background] Bedenko A.S. Metabolic factors in pathogenesis of migraine and unsteadiness. Medical alphabet. 2020;(33):18-20. (In Russ.) https://doi.org/10.33667/2078-5631-2020-33-18-20
- [Result] Bedenko A.S. Vertigo caused by vestibular migraine: current problems of pathogenesis, diagnostics and therapy. Epilepsy and paroxysmal conditions. 2020;12(3):177-181. (In Russ.)https://doi.org/10.17749/2077-8333/epi.par.con.2020.032